CLINICAL TRIAL: NCT05046743
Title: Intestinal Dysmotility in Patients With Functional Digestive Symptoms
Brief Title: Intestinal Dysmotility: Effect of Colonic Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PR(AG)56/2018B
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonic gas load (Experimental)
  Interventions: Other: Colonic gas load
- Sham (Sham Comparator)
  Interventions: Other: Sham load

INTERVENTIONS:
Other: Colonic gas load — Colonic infusion of gas via an anal cannula
  Arms: Colonic gas load
Other: Sham load — Sham infusion of gas via an anal cannula
  Arms: Sham

SUMMARY:
Abnormal motility patterns in the jejunum can be detected in patients with prominent colonic distension, and it is not clear whether these abnormalities reflect a primary jejunal dysfunction or are due to a reflex distortion. The aim of the study is to determine the effect of colonic filling on jejunal postprandial motility using high-resolution manometry.

Healthy subjects will be studied following a controlled, parallel, randomized, single-blind experimental design. On the study day, nutrients will be continuously infused in the proximal jejunum (2 Kcal/min) during a 2-h period to induce a steady-state postprandial motor pattern. Jejunal motility will be concomitantly recorded using a water-perfused, high-resolution manometry catheter. After 1 hour of postprandial recording (basal period), a gas mixture will be infused during 7.5 minutes via a rectal tube (720 mL or sham infusion), and jejunal motility will be recorded for another hour.

ELIGIBILITY:
Inclusion Criteria:

* No digestive symptoms

Exclusion Criteria:

* Organic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Small bowel contractility | 10 minutes
  Number of contractions

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No